CLINICAL TRIAL: NCT03517956
Title: A Multicenter Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of the Combination of Rogaratinib and Copanlisib in Patients With FGFR-positive, Locally Advanced or Metastatic Solid Tumors
Brief Title: Phase 1 Study of the Combination of Rogaratinib With Copanlisib in Patients With Fibroblast Growth Factor Receptor (FGFR)-Positive, Locally Advanced or Metastatic Solid Tumors
Acronym: ROCOCO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19774; 2018-000419-26 (EudraCT Number)
Record Dates: First submitted 2018-05-03; First posted 2018-05-08 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Advanced or Metastatic Solid Tumor
Keywords: Phase I; Locally advanced or metastatic solid tumor; Urothelial cancer; FGFR inhibitor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Rogaratinib; copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with FGFR1-4 - positive solid tumors (Experimental): Dose escalation:
  The starting dose of the combination will be escalated in a stepwise fashion, escalating one drug at a time.
  Dose expansion (urothelial cancer):
  Patients in the dose expansion will be treated with the combination identified in the dose escalation part of the study.
  Interventions: Drug: Rogaratinib (BAY1163877); Drug: Copanlisib (BAY80-6946)

INTERVENTIONS:
Drug: Rogaratinib (BAY1163877) — Dose escalation:
  Starting dose is rogaratinib 400 mg twice daily (b.i.d.) in continuous 28-day cycles from Cycle 1 Day 3 onwards.
  Dose expansion:
  With dose identified in dose escalation part.
Drug: Copanlisib (BAY80-6946) — Dose escalation:
  Starting dose is 45 mg on Days 1, 8 and 15 of each 28-day cycle.
  Dose expansion:
  With dose identified in dose escalation part.

SUMMARY:
The primary objective of this study is to determine the safety, tolerability, maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) and efficacy of rogaratinib in combination with copanlisib in patients with locally advanced or metastatic solid tumors that are mRNA-positive for at least one FGFR1-4 subtype.

The secondary objectives of this study are to characterize the pharmacokinetics (PK) of rogaratinib and copanlisib alone and in combination, and to assess the anti-tumor efficacy of rogaratinib in combination with copanlisib for locally advanced or metastatic solid tumors that are mRNA-positive for at least one FGFR1-4 subtype.

ELIGIBILITY:
Inclusion Criteria:

* High FGFR mRNA expression levels (RNAscope score of ≥3; measurement is part of this protocol) in archival or fresh tumor biopsy specimen.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
* At least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) in contrast enhanced (unless contraindicated) CT or MRI.
* Adequate bone marrow, liver and renal function.
* Glomerular filtration rate (GFR) ≥ 30 mL/min/1.73 m*2 according to the Modification of Diet in Renal Disease (MDRD) formula.
* Left ventricular ejection fraction (LVEF) equal to or above the lower limit of normal (LLN) at the institution.
* Life expectancy of at least 3 months.
* For the dose escalation part: Patients with histologically confirmed, locally advanced or metastatic solid tumors who are not candidates for or refuse standard therapy or whose disease progressed and for which standard anti-cancer treatment is no longer effective, excluding primary brain or spinal tumors. Patients who have been advised with all standard treatment options and still refuse them must be documented and can be allowed to enter the trial.
* For the dose expansion part: Patients with histologically confirmed, locally advanced or metastatic urothelial carcinoma (transitional cell carcinoma) including urinary bladder, renal pelvis, ureters, urethra who are not candidates for or refuse standard therapy or whose disease progressed and for which standard anticancer treatment is no longer effective. Patients who have been advised with all standard treatment options and still refuse them must be documented and can be allowed to enter the trial.

Exclusion Criteria:

* Previous or concurrent cancer that is distinct from tumor for which the patient is enrolled in the study, except

  * curatively treated cervical carcinoma in situ
  * treated basal-cell carcinoma
  * localized prostate cancer treated with curative intent and known absence of prostate-specific antigen (PSA) relapse or incidental prostate cancer (T1/T2a, Gleason score ≤ 6, and PSA ≤ 10 ng/mL undergoing active surveillance and treatment-naïve)
  * any cancer curatively treated > 3 years before planned start of study treatment.
* Ongoing or previous anti-cancer treatment within 4 weeks of study treatment start (or 6 weeks for mitomycin C, nitrosoureas and monoclonal antibodies); with exceptions.
* Prior toxicity to anti-FGFR-directed or anti-PI3K-directed therapies leading to treatment discontinuation (previous exposure is allowed in other circumstances). If prior toxicity to anti-FGFR-directed or anti-PI3K-directed therapies leading to treatment discontinuation is different from the known safety profile of rogaratinib or copanlisib, enrollment is allowed.
* Symptomatic brain or meningeal metastatic tumors unless the patient is >6 months from definitive therapy, has no evidence of tumor growth on an imaging study and is clinically stable with respect to the tumor at the start of study treatment. Also the patient must not be undergoing acute steroid therapy or taper (chronic steroid therapy is acceptable provided that the dose is stable for one month prior to and following screening radiographic studies).
* History or current condition of an uncontrolled cardiovascular disease including congestive heart failure NYHA > Class 2, unstable angina (symptoms of angina at rest) or new-onset angina (within last 3 months) or myocardial infarction within past 6 months and cardiac arrhythmias requiring anti-arrhythmic therapy (beta-blockers or digoxin are permitted).
* Active hepatitis B (HBV) or C (HCV) infection.
* Active clinically serious infections (≥ CTCAE v4.03 Grade 2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to 32 months
Incidence of drug-related TEAEs | Up to 32 months
Incidence of treatment-emergent serious adverse events (TESAEs) | Up to 32 months
Incidence of Dose-limiting toxicities (DLTs) | Approximately 10 months
Objective response rate (ORR) at recommended dose | Up to 32 months
  ORR in patients receiving the recommended dose of the rogaratinib-copanlisib-combination during the dose expansion part

SECONDARY OUTCOMES:
Maximum plasma concentration of Copanlisib (Cmax) | 0 (pre-dose), 0.5, 1 (end of infusion), 2, 4, 8, 24, 48 hours after drug administration (Days 1, 2, 3) and 0, 0.5, 1, 2, 4, 8, 24, 48 hours after drug administration (Days 15, 16, 17) in dose escalation
Area under the plasma concentration versus time curve of Copanlisib (AUC (0-48)) | 0 (pre-dose), 0.5, 1 (end of infusion), 2, 4, 8, 24, 48 hours after drug administration (Days 1, 2, 3) and 0, 0.5, 1, 2, 4, 8, 24, 48 hours after drug administration (Days 15, 16, 17) in dose escalation
Area under the plasma concentration versus time curve of Rogaratinib (AUC (0-8)) | 0 (pre-dose), 0.5, 1, 2, 4, 6, 8 hours after drug (Day 14) and 0 (pre-dose), 0.5, 1, 2, 4, 6, 8, 24, 48 hours after drug (Days 15 to 17) in dose escalation; 0 (pre-dose) and 1 hour after drug on Day 1 of dose expansion
Maximum plasma concentration of Rogaratinib (Cmax) | 0 (pre-dose), 0.5, 1, 2, 4, 6, 8 hours after drug (Day 14) and 0 (pre-dose), 0.5, 1, 2, 4, 6, 8, 24, 48 hours after drug (Days 15 to 17) in dose escalation; 0 (pre-dose) and 1 hour after drug on Day 1 of dose expansion
Objective response rate (ORR) | Up to 32 months
Disease control rate (DCR) | Up to 32 months
Duration of response (DOR) for Partial Response and Complete Response | Up to 32 months
Progression-free survival (PFS) | Up to 32 months
Overall survival (OS) | Up to 32 months

CONTACTS AND LOCATIONS:
Locations (20):
- United States (7):
  - USC Norris Hospital and Clinics, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute - Detroit, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Tyler Cancer Center, Tyler, Texas
- Belgium (3):
  - CU Saint-Luc/UZ St-Luc, Bruxelles - Brussel
  - UZ Antwerpen, Edegem
  - CHU de Liège, Liège
- Germany (3):
  - Krankenhaus Nordwest, Frankfurt am Main, Hesse
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Klinikum der Universität Würzburg, Würzburg
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Center Singapore, Singapore
- South Korea (3):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (2):
  - Ciutat Sanitària i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.